CLINICAL TRIAL: NCT06781138
Title: Comparison Between Conventional Versus 3D-Designed and Printed Stabilization Splints for Treatment of TMD Patients: A Randomized Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdallah Ahmed Hassan, Resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2461994
Record Dates: First submitted 2025-01-14; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Temporomandibular Disorders (TMD)
Keywords: TMD Joint
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional stabilization splint (Active Comparator)
  Interventions: Device: Conventional stabilization splint
- 3D designed and printed stabilization splint (Experimental)
  Interventions: Device: 3D designed and printed stabilization splints

INTERVENTIONS:
Device: Conventional stabilization splint — conventional versus 3D designed and printed stabilization splints
  Arms: Conventional stabilization splint
Device: 3D designed and printed stabilization splints — Conventional versus 3D designed and printed stabilization splints
  Arms: 3D designed and printed stabilization splint

SUMMARY:
This study is a randomized clinical trial comparing the effectiveness of conventional stabilization splints versus 3D-designed and printed stabilization splints in treating temporomandibular disorders (TMDs). TMD is a common cause of orofacial pain affecting the jaw joint and surrounding muscles. The trial evaluates outcomes such as pain reduction, clinical improvement, patient satisfaction, and time efficiency. By exploring a fully digital workflow for splint fabrication, this study aims to provide evidence on whether the newer 3D-printed approach offers superior results to conventional methods in terms of clinical effectiveness and procedural efficiency.

DETAILED DESCRIPTION:
This study is a randomized clinical trial designed to evaluate the efficacy of 3D-designed and printed stabilization splints compared to conventional stabilization splints in managing temporomandibular disorders (TMDs) of muscular origin. TMD is a prevalent orofacial condition characterized by pain and dysfunction in the temporomandibular joint (TMJ) and associated structures, significantly impacting patients' quality of life. Stabilization splints are a widely used conservative treatment for TMD, aiming to alleviate symptoms by stabilizing occlusion, reducing parafunctional habits, and promoting muscle relaxation. Despite their popularity, controversies remain about their optimal design and long-term efficacy, especially with recent advancements in digital fabrication technologies.

Study Objectives The primary aim is to assess whether 3D-designed and printed stabilization splints offer superior clinical outcomes compared to conventional splints. Outcomes include pain reduction (measured using the Visual Analog Scale, VAS) and clinical improvement based on Diagnostic Criteria for TMD (DC/TMD) evaluations. Secondary objectives include measuring patient satisfaction, chairside time during splint fabrication, and changes in maximal unassisted incisal opening.

Study Design This is a single-blinded, randomized, parallel-group clinical trial with a 1:1 allocation ratio. The study will be conducted at the outpatient clinic of the Department of Orthodontics, Faculty of Dentistry, Cairo University. Adult patients aged 18-40 with muscular TMD are eligible, provided they meet inclusion criteria and have no prior orthodontic treatments.

Methodology

Participants will be randomly assigned to one of two groups:

Intervention Group: Patients will undergo direct intraoral scanning using a digital scanner. The data will be used to design and fabricate stabilization splints using a fully digital, 3D-printing workflow.

Comparator Group: Patients will have conventional alginate impressions taken. Stabilization splints will be fabricated using cold-cure acrylic resin.

Patients in both groups will be instructed to wear their splints at night only. Follow-up assessments will occur at 2, 4, 8, and 12 weeks to evaluate outcomes.

12) Outcomes:

Primary:

• Measuring clinical improvement and pain level using VAS

Secondary:

* Measuring the patient satisfaction during wearing of the splint using VAS
* Chairside time taken during conventional splint impression and fabrication vs digital splint intraoral scan and design
* Changes in maximal incisal opening (fitting day/8 weeks) Significance This study addresses an important clinical question by comparing traditional and modern techniques for splint fabrication. By leveraging a digital workflow, it aims to provide insights into whether 3D-printed splints can improve clinical outcomes, enhance patient satisfaction, and reduce the time required for fabrication, potentially advancing TMD management practices.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged (18-40) presenting with myalgia.

Exclusion Criteria:

* Previous orthodontic treatment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
clinical improvement | after 8 weeks
  Visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah Ahmed Hassan Hamed Refai, MSc candidate, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided